CLINICAL TRIAL: NCT05036733
Title: Effects of IL-4R-alpha Inhibition (Dupixent) Inhibition On The Respiratory Microbiome And Immunologic Correlates In Patients With Severe Asthma
Brief Title: Effects of Interleukin (IL)- 4R-alpha Inhibition on Respiratory Microbiome and Immunologic Correlates in Severe Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Yvonne J Huang, Associate Professor of Internal Medicine and Microbiology/Immunology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00196809
Record Dates: First submitted 2021-08-30; First posted 2021-09-08 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Asthma
Keywords: Inhaled corticosteroids; Dupilumab
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dupilumab (Experimental)
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Participants will receive 8 doses of Dupilumab. The initial loading dose (visit 1) of 600 milligrams (two 300 milligram injections) will be given subcutaneously (SQ). Then the participants will receive 300 milligrams SQ every other week (q 2 weeks) either at a study visit or self-administered at home between visits.
  Additionally, participants will complete questionnaires, have specimens collected, as well as perform breathing procedures at various timepoints.
  Other Names: Dupixent

SUMMARY:
The overall goal of this study is to understand biological responses related to dupilumab treatment among severe asthma patients.

Not all asthma is the same, and characteristics of asthma vary from person to person. The study will investigate whether the study drug can help to improve the health of participants lungs, boost immune response, as well as improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed/managed severe asthma patients that are clinically eligible for dupilumab
* Current treatment with a medium-to-high-dose inhaled glucocorticoid (fluticasone propionate at a total daily dose of greater or equal (≥) 440 μg or equipotent equivalent) plus up to at least one additional controller (e.g., a long-acting β2-agonist or leukotriene receptor antagonist)
* Eosinophilic asthma phenotype (blood eosinophil level >300) or asthma requiring daily oral corticosteroids
* Asthma that is uncontrolled, as defined by a score on the Asthma Control Test of 19 or lower, or a worsening of asthma in the past year that led to an asthma hospitalization, Emergency Department visit, or 3 days of oral corticosteroids
* Severity of asthma that, in the opinion of the subject's asthma care specialist, requires dupilumab for control
* For women of childbearing age: agree to use birth control or remain abstinent during the duration of the study.

Exclusion Criteria:

* Patients with diagnosis of other chronic lung diseases (e.g. Chronic obstructive pulmonary disease (COPD), idiopathic pulmonary fibrosis, Churg-Strauss syndrome, Allergic bronchopulmonary aspergillosis, etc.)
* Current smoker or reported smoking within 1 month of the screening visit (tobacco or any inhaled recreational product)
* Greater than 10 total pack-year of cigarette smoking history
* Treatment with oral corticosteroids for an asthma exacerbation 1 month prior to screening or during the screening period
* Use of any biologic therapy for asthma within the past 3 months
* Respiratory or Gastrointestinal illness within 1 month prior to screening or during the screening period
* Treatment with antibiotics for acute infections within six weeks prior to screening or during the screening period.
* Pregnancy at enrollment or during the study
* Known hypersensitivity to dupilumab or its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Huang, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dupilumab
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dupilumab
Number analyzed (Participants) | 15
Age, Continuous [Median (Standard Deviation); unit: years] | 59 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14
  Race other than White | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
FEV1:FVC [Median (Standard Deviation); unit: ratio] | 0.75 (0.12)
Body-mass index [Median (Standard Deviation); unit: (kg/m^2)] | 30.1 (12.7)
Fractional exhaled nitric oxide (FeNO) [Median (Standard Deviation); unit: parts per billion] | 32 (33)
Asthma Control Test (ACT) score [Median (Standard Deviation); unit: score on a scale] — The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control.
  score on a scale | 15 (5)
Sino-nasal outcome test (SNOT-22) score [Median (Standard Deviation); unit: score on a scale] — The possible range of Total SNOT scores is between 0 to 110 for the SNOT-22.
  Higher scores indicate greater rhinosinusitis-related health burden.
  score on a scale | 44 (16)
mini-Asthma Quality of Life Questionnaire (mAQLQ) score [Median (Standard Deviation); unit: score on a scale] — This is a patient self-administered questionnaire with 15 questions covering 4 domains: Symptoms (5 questions), Activity Limitations (4 questions), Emotional Function (3 questions), and Environmental Stimuli (3 questions). Scores range from 0-6 (lower is worse). The mini AQLQ score is calculated as the average of domain items. The minimum clinically important difference is 0.5.
  Overall score (average of 15 questions): add up responses to all questions, and divide by 15.
  score on a scale | 4.2 (1.2)
alpha-diversity of respiratory (sputum) microbiota: Shannon index [Mean (Standard Deviation); unit: Shannon's index] — α-diversity was calculated using the Shannon Diversity Index at the species level from induced sputum samples. A higher Shannon Diversity Index value indicates higher diversity.
  Shannon's index | 3.08 (0.36)
Relative abundances of respiratory (sputum) microbiota members [Mean (Standard Deviation); unit: percentages] — Relative abundance was calculated by finding the proportion of a classified species out of all bacterial classifications in an induced sputum sample.
  percentages
    Streptococcus salivarius | 17.8 (14.5)
    Streptococcus sanguinis | 2.2 (1.2)
    Streptococcus parasanguinis | 10.8 (8.4)
    Bifidobacterium longum | 0.81 (1.5)
    Tropheryma whipplei | 2.23 (2.4)
    Bifidobacterium dentium | 0.55 (0.8)
    Streptococcus gordonii | 2.9 (3.7)
    Parvimonas micra | 3.5 (4.5)
    Streptococcus anginosus | 3.5 (8.7)
    Rothia mucilaginosa | 7.2 (5.6)
Respiratory bacterial burden (#bacterial cells, sputum) [Mean (Standard Deviation); unit: bacterial cells] | 4,622,000,000 (6,443,000,000)
alpha-diversity of stool microbiota: Shannon index [Mean (Standard Deviation); unit: score on a scale] — α-diversity was calculated using the Shannon diversity Index at the species level from stool samples. A higher Shannon Diversity Index value indicates higher diversity.
  score on a scale | 3.20 (0.31)
Oral Corticosteroid Use [Count of Participants; unit: Participants] — Number of participants using oral corticosteroids
  Participants | 1
Blood eosinophils [Mean (Standard Deviation); unit: cells/microliter] | 200 (200)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Alpha-diversity of Respiratory Microbiota
Description: α-diversity was calculated using the Shannon Diversity Index at the species level from induced sputum samples obtained at Baseline and after 1 month on dupilumab. The change in diversity was calculated by aggregating all participants' calculated diversity and then finding the difference between time points. A higher Shannon Diversity Index value indicates higher diversity. A value of zero indicates the presence of only one kind of species of bacteria.
Time Frame: Baseline (before dupilumab), 1 month
Population: While 15 participants completed treatment, not all participants were able to provide biosamples. All data collected from available samples is provided here.
Measure: Mean (Standard Deviation); unit: Shannon's index
Arm/Group | Dupilumab
Number analyzed (Participants) | 7
Shannon's index | 0.13 (0.29)

2. Primary Outcome: Changes in Alpha-diversity of Respiratory Microbiota
Description: α-diversity was calculated using the Shannon Diversity Index at the species level from induced sputum samples obtained at baseline and after 4 months on dupilumab. The change in diversity was calculated by aggregating all participants' calculated diversity and then finding the difference between time points. A higher Shannon Diversity Index value indicates higher diversity. A value of zero indicates the presence of only one kind of species of bacteria.
Time Frame: Baseline (before dupilumab), 4 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Shannon's index
Arm/Group | Dupilumab
Number analyzed (Participants) | 7
Shannon's index | 0.14 (0.30)

3. Primary Outcome: Changes in Alpha-diversity of Respiratory Microbiota
Description: α-diversity was calculated using the Shannon Diversity Index at the species level from induced sputum samples obtained after 1 month and after 4 months on dupilumab. The change in diversity was calculated by aggregating all participants' calculated diversity and then finding the difference between time points. A higher Shannon Diversity Index value indicates higher diversity. A value of zero indicates the presence of only one kind of species of bacteria.
Time Frame: 1 month, 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Shannon's index
Arm/Group | Dupilumab
Number analyzed (Participants) | 6
Shannon's index | -0.09 (0.41)

4. Primary Outcome: Change in Beta-diversity of Respiratory Microbiota
Description: Beta-diversity was calculated using the Bray-Curtis Distance at the species level from induced sputum samples obtained at baseline and after 1 month on dupilumab. The change in diversity was calculated by aggregating all participants' distance between time points. Bray-Curtis dissimilarity ranges from 0 to 1. A higher Bray-Curtis Distance, which is unitless, indicates a greater difference in diversity between the time points.
Time Frame: Baseline (before dupilumab), 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 7
score on a scale | .82 (0.17)

5. Primary Outcome: Change in Beta-diversity of Respiratory Microbiota
Description: Beta-diversity was calculated using the Bray-Curtis Distance at the species level from induced sputum samples obtained at baseline and after 4 months on dupilumab. The change in diversity was calculated by aggregating all participants' distance between time points. Bray-Curtis dissimilarity ranges from 0 to 1. A higher Bray-Curtis Distance indicates a greater difference in diversity between time points.
Time Frame: Baseline (before dupilumab), 4 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 7
score on a scale | 0.82 (0.17)

6. Primary Outcome: Change in Beta-diversity of Respiratory Microbiota
Description: Beta-diversity was calculated using the Bray-Curtis Distance at the species level from induced sputum samples obtained after 1 month and after 4 months on dupilumab. The change in diversity was calculated by aggregating all participants' distance between time points. Bray-Curtis dissimilarity ranges from 0 to 1. A higher Bray-Curtis Distance indicates a greater difference in diversity between time points.
Time Frame: 1 month, 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 6
score on a scale | 0.81 (0.19)

7. Primary Outcome: Change in Relative Abundances of Microbiota Members
Description: Relative abundance was calculated by finding the proportion of a classified species out of all bacterial classifications in an induced sputum sample. Relative abundance was calculated at baseline and after 1 month on dupilumab. The change in relative abundance of each species across all available samples was calculated by taking the difference between time points.
Time Frame: Baseline (before dupilumab), 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of bacterial classification
Arm/Group | Dupilumab
Number analyzed (Participants) | 7
percentage of bacterial classification
  Streptococcus salivarius | -5.9 (0.09)
  Streptococcus sanguinis | -2.4 (0.04)
  Streptococcus parasanguinis | 0.03 (0.05)
  Bifidobacterium longum | 0.03 (0.02)
  Tropheryma whipplei | 0.2 (0.04)
  Bifidobacterium dentium | 0.3 (0.01)
  Streptococcus gordonii | 1.0 (0.02)
  Parvimonas micra | 1.6 (0.04)
  Streptococcus anginosus | 1.6 (0.04)
  Rothia mucilaginosa | 2.0 (0.05)

8. Primary Outcome: Change in Relative Abundances of Microbiota Members
Description: Relative abundance was calculated by finding the proportion of a classified species out of all bacterial classifications in an induced sputum sample. Relative abundance was calculated at baseline and after 4 months on dupilumab. The change in relative abundance of each species across all available samples was calculated by taking the difference between time points.
Time Frame: Baseline (before dupilumab), 4 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of bacterial classification
Arm/Group | Dupilumab
Number analyzed (Participants) | 7
percent of bacterial classification
  Streptococcus salivarius | -0.2 (0.07)
  Streptococcus sanguinis | 1.1 (0.02)
  Streptococcus parasanguinis | -2.6 (0.1)
  Bifidobacterium longum | -1.6 (0.04)
  Tropheryma whipplei | 2.4 (0.03)
  Bifidobacterium dentium | -3.1 (0.07)
  Streptococcus gordonii | 0.05 (0.03)
  Parvimonas micra | 0.6 (0.04)
  Streptococcus anginosus | 1.1 (0.04)
  Rothia mucilaginosa | -4.0 (0.09)

9. Primary Outcome: Change in Relative Abundances of Microbiota Members
Description: Relative abundance was calculated by finding the proportion of a classified species out of all bacterial classifications in an induced sputum sample. Relative abundance was calculated after 1 month and after 4 months on dupilumab. The change in relative abundance of each species across all available samples was calculated by taking the difference between time points.
Time Frame: 1 month, 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of bacterial classification
Arm/Group | Dupilumab
Number analyzed (Participants) | 6
percent of bacterial classification
  Streptococcus salivarius | 8.3 (0.1)
  Streptococcus sanguinis | 3.3 (0.04)
  Streptococcus parasanguinis | -3.5 (0.12)
  Bifidobacterium longum | -1.6 (0.02)
  Tropheryma whipplei | 0.1 (0)
  Bifidobacterium dentium | -4.5 (0.08)
  Streptococcus gordonii | -1.6 (0.04)
  Parvimonas micra | -1.2 (0.02)
  Streptococcus anginosus | -0.5 (0.01)
  Rothia mucilaginosa | -2.0 (0.05)

10. Primary Outcome: Change in Respiratory Bacterial Burden
Description: Bacterial burden was estimated by scaling species relative abundances to a known cell count of Imtechella halotolerans (Zymo) that was spiked into an induced sputum sample before extraction for sequencing. Bacterial burden was calculated at baseline and after 1 month on dupilumab. The change in bacterial burden was calculated by aggregating all burden values per participant and taking the difference between time points.
Time Frame: Baseline (before dupilumab), 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Dupilumab
Number analyzed (Participants) | 7
cells | -16,117,353,849 (19,829,305,914)

11. Primary Outcome: Change in Respiratory Bacterial Burden
Description: Bacterial burden was estimated by scaling all species relative abundances to a known cell count of Imtechella halotolerans that was spiked into sputum samples before extraction for sequencing. Bacterial burden was calculated at baseline and after 4 months on dupilumab. The change in bacterial burden was calculated by aggregating all burden values per participant and taking the difference between time points.
Time Frame: Baseline (before dupilumab), 4 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Dupilumab
Number analyzed (Participants) | 7
cells | -25,294,991,477 (44,588,805,244)

12. Primary Outcome: Change in Respiratory Bacterial Burden
Description: Bacterial Burden was estimated by scaling the species relative abundance to a known cell count of I. Halotolerans that was spiked into an induced sputum sample before extraction for sequencing. Bacterial burden was calculated at after 1 month and after 4 months on dupilumab. The change in bacterial burden was calculated by aggregating all burden values per participant and taking the difference between time points.
Time Frame: 1 month, 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Dupilumab
Number analyzed (Participants) | 6
cells | -9,927,388,331 (44,588,805,244)

13. Primary Outcome: Changes in Alpha-diversity of Stool Microbiota
Description: α-diversity was calculated using the Shannon diversity index at the species level from stool samples obtained at baseline and after 1 month on dupilumab. The change in diversity was calculated by aggregating all participants' calculated diversity and then finding the difference between time points. A higher Shannon Diversity Index value indicates higher diversity. A value of zero indicates the presence of only one kind of species of bacteria.
Time Frame: Baseline (before dupilumab), 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Shannon's index
Arm/Group | Dupilumab
Number analyzed (Participants) | 4
Shannon's index | 0.07 (0.24)

14. Primary Outcome: Changes in Alpha-diversity of Stool Microbiota
Description: α-diversity was calculated using the Shannon diversity Index at the species level from stool samples obtained at baseline and after 4 months on dupilumab. The change in diversity was calculated by aggregating all participants' calculated diversity and then finding the difference between time points. A higher Shannon Diversity Index value indicates higher diversity. A value of zero indicates the presence of only one kind of species of bacteria.
Time Frame: Baseline (before dupilumab), 4 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Shannon's index
Arm/Group | Dupilumab
Number analyzed (Participants) | 3
Shannon's index | 0.04 (0.29)

15. Primary Outcome: Changes in Alpha-diversity of Stool Microbiota
Description: α-diversity was calculated using the Shannon Diversity Index at the species level from stool samples. Shannon's Diversity Index values were obtained after 1 month and after 4 months on dupilumab. The change in diversity was calculated by aggregating all participants' calculated diversity and then finding the difference between time points. A higher Shannon Diversity Index value indicates higher diversity. A value of zero indicates the presence of only one kind of species of bacteria.
Time Frame: 1 month, 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Shannon's index
Arm/Group | Dupilumab
Number analyzed (Participants) | 2
Shannon's index | 0.42 (0.67)

16. Primary Outcome: Change in Beta-diversity of Stool Microbiota
Description: Beta-diversity was calculated using the Bray-Curtis Distance at the species level from stool samples. Samples were obtained baseline and after 1 month on dupilumab and the Bray-Curtis Distance calculated. The change in diversity was calculated by aggregating all participants' distance between time points. Bray-Curtis dissimilarity ranges from 0 to 1. A higher Bray-Curtis Distance indicates a greater difference in diversity between time points..
Time Frame: Baseline (before dupilumab), 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 4
score on a scale | 0.72 (0.14)

17. Primary Outcome: Change in Beta-diversity of Stool Microbiota
Description: Beta-diversity was calculated using the Bray-Curtis Distance at the species level from stool samples obtained at baseline and after 4 months on dupilumab. The change in diversity was calculated by aggregating all participants' distance between time points. Bray-Curtis dissimilarity ranges from 0 to 1. A higher Bray-Curtis Distance indicates a greater difference in diversity between time points.
Time Frame: Baseline (before dupilumab), 4 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 3
score on a scale | 0.75 (0.12)

18. Primary Outcome: Change in Beta-diversity of Stool Microbiota
Description: Beta-diversity was calculated using the Bray-Curtis Distance at the species level from stool samples obtained after 1 month and after 4 months on dupilumab. The change in diversity was calculated by aggregating all participants' distance between time points. Bray-Curtis dissimilarity ranges from 0 to 1. A higher Bray-Curtis Distance indicates a greater difference in diversity between time points.
Time Frame: 1 month, 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 2
score on a scale | 0.71 (0.14)

19. Secondary Outcome: Forced Expiratory Volume ( FEV1) / Forced Vital Capacity (FVC) Ratio
Description: Ratio of the volume of air exhaled in 1 sec (FEV1) divided by the total volume exhaled (FVC). FEV1/FVC < 0.70 (or less than lower limit of age-predicted normal) is clinically diagnostic of obstructive lung disease.
Time Frame: Baseline, 1 month, 4 months
Measure: Median (Full Range); unit: ratio
Arm/Group | Dupilumab
Number analyzed (Participants) | 15
ratio
  Visit 1 | 0.75 [0.53 to 0.91]
  Visit 2 | 0.78 [0.51 to 0.93]
  Visit 3 | 0.77 [0.54 to 0.92]

20. Secondary Outcome: Forced Expiratory Volume (FEV1)
Description: FEV1 measure reported as a percentage of predicted FEV1.
Time Frame: Baseline, 1 month, 4 months
Measure: Median (Full Range); unit: percent of predicted volume
Arm/Group | Dupilumab
Number analyzed (Participants) | 15
percent of predicted volume
  Visit 1 | 85 [54 to 120]
  Visit 2 | 88 [61 to 137]
  Visit 3 | 89 [57 to 128]

21. Secondary Outcome: Change in Fractional Exhaled Nitric Oxide (FeNO)
Description: Fractional exhaled nitric oxide is a clinical biomarker for type 2 airway inflammation. FeNO >25 is considered indicative of type 2 airway inflammation.
Time Frame: Baseline, 1 month, 4 months
Measure: Median (Full Range); unit: parts per billion
Arm/Group | Dupilumab
Number analyzed (Participants) | 15
parts per billion
  Visit 1 | 32 [5 to 127]
  Visit 2 | 24 [6 to 42]
  Visit 3 | 17 [5 to 45]

22. Secondary Outcome: Asthma Control Test (ACT)
Description: The Asthma Control Test is a clinically validated questionnaire that assesses level of asthma control based on a 4-week recall of symptoms and daily functioning captured in 5 items. Each item is scored on a 5-point scale, and the total score is the sum of the values for all 5 items (range 5-25). A score of 5 represents worst-controlled asthma and 25 represents best-controlled asthma. An ACT score >19 indicates well-controlled asthma; the minimal clinically important difference in score is 3.
Time Frame: Baseline, 1 month, 4 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 15
score on a scale
  Visit 1 | 15 [7 to 21]
  Visit 2 | 21 [9 to 25]
  Visit 3 | 21 [11 to 25]

23. Secondary Outcome: Mini Asthma Quality of Life Questionnaire Score (mAQLQ)
Description: The mini-Asthma Quality of Life Questionnaire (mAQLQ) consists of 15 questions covering 4 domains: symptoms (5 questions), activity limitations (4 questions), emotional function (3 questions), and environmental stimuli (3 questions). The recall time for the mAQLQ is 2 weeks and each item is scored on a 7-point scale. Total scores per participant are the average of the 15 items and range from 1-7, with higher scores indicative of better quality of life. The minimum clinically important difference is 0.5.
Time Frame: Baseline, 1 month, 4 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 15
score on a scale
  Visit 1 | 4.2 [1.9 to 7.0]
  Visit 2 | 5.2 [2.7 to 7.0]
  Visit 3 | 5.6 [3.5 to 6.9]

24. Secondary Outcome: Sino-nasal Outcome Test (SNOT-22)
Description: This is a 22 item questionnaire. Each item is rated as follows: 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be. The score ranges between 0 and 110. A higher score means worse outcome.
Time Frame: Baseline, 1 month, 4 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 15
score on a scale
  Visit 1 | 44 [3 to 58]
  Visit 2 | 24 [1 to 63]
  Visit 3 | 21 [5 to 56]

25. Secondary Outcome: Change in Prescribed Maintenance Corticosteroid Use (Inhaled or Oral), Between Baseline and 4 Months.
Description: Count of participants whose maintenance corticosteroid prescription changed between baseline and 4 months.
Time Frame: Baseline, 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 15
Participants | 0

26. Secondary Outcome: Number of Asthma Exacerbations Requiring at Least 3 Days of Oral Corticosteroids
Description: Number of asthma exacerbations requiring at least 3 days of oral corticosteroids across the entire study population over the course of the study.
Time Frame: up to 4 months
Measure: Number; unit: count of exacerbations
Arm/Group | Dupilumab
Number analyzed (Participants) | 15
count of exacerbations | 1

ADVERSE EVENTS:
Time Frame: 4 months
Description: Non-serious adverse event information was not collected.
Arm/Group | Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab (N=15)
Pneumonia-attributed acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory difficulty requiring hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute myeloid leukemia diagnosis (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT05036733/Prot_SAP_000.pdf